CLINICAL TRIAL: NCT00414427
Title: Using Ultrasonography to Predict Clinical Response to Intraarticular Corticosteroids in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Kenneth Kalunian, M.D., Professor of Medicine, UCSD
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 051420
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2006-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Ultrasonography; Corticosteroids
MeSH Terms: conditions — Osteoarthritis, Knee

INTERVENTIONS:
Procedure: Intraarticular steroids

SUMMARY:
The primary purposes of this study are the following:

1. To evaluate whether the presence of inflammatory knee osteoarthritis as determined by ultrasonography can be used as a clinical predictor of patient response to intra-articular corticosteroids.
2. To prospectively evaluate clinical responsiveness of intraarticular corticosteroids with the inflammatory phenotype of knee OA using a randomized, placebo controlled clinical design.
3. To evaluate whether lower extremity strength is improved with intraarticular corticosteroid injection.

The investigators hypothesize that patients with signs of inflammation by ultrasonography such as synovitis and effusion will respond better to intraarticular corticosteroid injection.

DETAILED DESCRIPTION:
Osteoarthritis (OA) has previously been thought to be a non-inflammatory condition whose pathologic hallmark is destruction of hyaline cartilage. It is now realized that OA results from a complex interplay of multiple factors, including local inflammatory processes. Evidence suggests that synovitis which is the usual presenting sign of inflammatory arthritis is also frequently present in OA.

The presence of inflammation in knee OA may explain why intra-articular (IA) corticosteroid injections have been shown to result in clinically and statistically significant reduction in osteoarthritic knee pain. Randomized controlled trials have shown that treated patients were less likely to have continuing pain and had significantly lower scores on a visual analogue scale (VAS) for pain. However, studies have failed to determine clinical predictors of response to IA steroid injection, including traditional indices of inflammation (heat, fluid, stiffness). One possibility is that local corticosteroids do no act to relieve pain by reducing synovitis. These putative mechanisms have yet to be elucidated. Perhaps a more plausible explanation is that current methods of assessing local inflammation in OA are inadequate.

Recent studies involving ultrasonography (US) demonstrate that US is a valid and reproducible tool for the detection of synovitis in the knee. It has been shown to be more sensitive than clinical examination and is relatively inexpensive and noninvasive.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients are eligible for the study if they are between 40 and 80 years old, have symptomatic knee OA requiring treatment, and have not responded adequately to treatment with acetominophen or NSAIDs.

Exclusion Criteria:

* Severe OA as defined by radiographic Kellgren and Lawrence Grade IV
* The patient being wheel-chair bound
* Previous knee operation on the affected side within the past year or history of total knee arthroplasty (affected side)
* Any IA steroid or injections in the last 3 months or viscosupplementation in the last 6 months
* Local sepsis
* Local skin conditions
* Serious concomitant medical illness.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To evaluate whether the presence of inflammatory knee osteoarthritis as determined by ultrasonography can be used as a clinical predictor of patient response to intra-articular corticosteroids.
To prospectively evaluate clinical responsiveness of intraarticular corticosteroids with the inflammatory phenotype of knee OA using a randomized, placebo controlled clinical design.

SECONDARY OUTCOMES:
To evaluate whether lower extremity strength is improved with intraarticular corticosteroid injection.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kalunian, M.D., Principal Investigator — Univeristy of California at San Diego
Locations (2):
- United States (2):
  - Thorton Hospital, La Jolla, California
  - La Jolla Veterans Affairs Medical Center, San Diego, California

REFERENCES:
- [Background] Godwin M, Dawes M. Intra-articular steroid injections for painful knees. Systematic review with meta-analysis. Can Fam Physician. 2004 Feb;50:241-8. PMID 15000335
- [Background] Gaffney K, Ledingham J, Perry JD. Intra-articular triamcinolone hexacetonide in knee osteoarthritis: factors influencing the clinical response. Ann Rheum Dis. 1995 May;54(5):379-81. doi: 10.1136/ard.54.5.379. PMID 7794044
- [Background] Walther M, Harms H, Krenn V, Radke S, Faehndrich TP, Gohlke F. Correlation of power Doppler sonography with vascularity of the synovial tissue of the knee joint in patients with osteoarthritis and rheumatoid arthritis. Arthritis Rheum. 2001 Feb;44(2):331-8. doi: 10.1002/1529-0131(200102)44:23.0.CO;2-0. PMID 11229463
- [Background] Karim Z, Wakefield RJ, Quinn M, Conaghan PG, Brown AK, Veale DJ, O'Connor P, Reece R, Emery P. Validation and reproducibility of ultrasonography in the detection of synovitis in the knee: a comparison with arthroscopy and clinical examination. Arthritis Rheum. 2004 Feb;50(2):387-94. doi: 10.1002/art.20054. PMID 14872480
- [Background] Jones A, Doherty M. Intra-articular corticosteroids are effective in osteoarthritis but there are no clinical predictors of response. Ann Rheum Dis. 1996 Nov;55(11):829-32. doi: 10.1136/ard.55.11.829. PMID 8976640